CLINICAL TRIAL: NCT05030181
Title: Efficacy of Kinesiology Tape Versus Postural Correction Exercises on Neck Disability in Nonspesific Nek Pain: A Randomized Single Blinded Clinical Trial
Brief Title: Efficacy of Kinesiology Tape on Neck Disability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Physical Medicine Rehabilitation Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Cansin Medin, principal investigator, Istanbul Physical Medicine Rehabilitation Training and Research Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: KAEK/2021.03.87
Record Dates: First submitted 2021-07-13; First posted 2021-09-01 (Actual); Last update posted 2021-09-22 (Actual); Status verified 2021-09

CONDITIONS: Pain; Myofascial Pain Syndrome; Trigger Point Pain, Myofascial
MeSH Terms: conditions — Pain; Myofascial Pain Syndromes | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: single blinded randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- kinesiotaping and exercise (Active Comparator): 'I'' strip kinesiotape will be applied with the space correction technique for the upper trapezius muscle, for a total of 4 sessions, 2 days a week, and the patients will be included in the 1-month home exercise program.
  Interventions: Other: kinesiotaping and exercise
- exercise (Active Comparator): 1-month home exercise program.
  Interventions: Other: exercise

INTERVENTIONS:
Other: kinesiotaping and exercise — kinesiotaping group, ''I'' strip kinesiotape will be applied with the space correction technique for the upper trapezius muscle, for a total of 4 sessions, 2 days a week, and the patients will be included in the 1-month home exercise program.
  Arms: kinesiotaping and exercise
Other: exercise — exercise
  Arms: exercise

SUMMARY:
Sixty participants with nonspecific neck pain were randomly assigned to either the kinesiotaping (n=30) or exercise (n=30) group.

At the beginning, at the 2nd week and at the 1st month, activity and rest pain with visual analog scale, cervical lateral flexion and rotation with goniometer, neck disability scale and trapezius thickness, trigger point volume, trigger point diameter, trigger point area (with ultrasonograpic imaging) will be evaluated.

After the initial evaluation of the patients in the kinesiotaping group, 'I' strip kinesiotape will be applied with the space correction technique for the upper trapezius muscle, for a total of 4 sessions, 2 days a week, and the patients will be included in the 1-month home exercise program. Patients will be evaluated at the start of treatment, Week 2, and Month.

Patients in the control group will only be included in the 1-month home exercise program. Patients will be evaluated at the start of treatment, Week 2, and Month 1.

The participants inclusion criteria were; age between 18 and 65 years, symptom duration of at least 3 months. The exclusion criteria were as follows: (1) a diagnosis of cervical radiculopathy or myelopathy, (2) a history of acute neck injury or cervical surgery (3) diagnosis of psychiatric disorders (4) recent trigger-point injection or participation in a physical treatment program witin the last 6 monhts (5) any allergies to the tape and (6) having already received treatment with kinesio-taping.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 65 years
* symptom duration of at least 3 months

Exclusion Criteria:

* a diagnosis of cervical radiculopathy or myelopathy
* a history of acute neck injury or cervical surgery
* diagnosis of psychiatric disorders
* recent trigger-point injection or participation in a physical treatment program witin the last 6 monhts
* any allergies to the tape and
* having already received treatment with kinesio-taping.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-06-05 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
visual analog scale | Baseline
  activity and rest pain with visual analog scale '0' no pain '10' severe pain
visual analog scale | 2nd week
  activity and rest pain with visual analog scale. '0' no pain '10' severe pain
visual analog scale | 1st month
  activity and rest pain with visual analog scale '0' no pain '10' severe pain

CONTACTS AND LOCATIONS:
Overall Officials: cansın m ceylan, Principal Investigator — istanbul physical medicine and rehabilitation research and training hospital
Locations (1):
- Cansın Medin Ceylan, Istanbul, None Selected, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No